CLINICAL TRIAL: NCT04172298
Title: The Study on the Relationship Among Meridian, Acupoint and Internal Visceral Organs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Basic Science
Other Study IDs: CMUH106-REC1-089
Record Dates: First submitted 2019-11-15; First posted 2019-11-21 (Actual); Last update posted 2019-11-21 (Actual); Status verified 2019-11

CONDITIONS: Meridian
Keywords: Meridian; Internal visceral organs; Zusanli; Shaohai; Acupoint

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- sham electroacupuncture (EA) session (Placebo Comparator): The stainless steels acupuncture needles inserted into the subcutaneous layer of Zusanli (cathode) and Shangjuxu acupints (anion) , and the needles connected to EA stimulator, but no electric discharge for 30 min.
  Interventions: Other: sham electroacupuncture (EA) session
- Zusanli session (Experimental): The acupuncture needles inserted into Zusanli (cathode) and Shangjuxu acupoints (anion), and twisting obtain qi, and the needles then connected to EA stimulator, the frequency was 2 Hz, the duration was 30 min, and the intensity was visual slightly muscle contraction.
  Interventions: Other: Zusanli session
- Shaohai session (Experimental): The methods were identical Zusanli group, but Shaohai acupoint (cathode), and 3 cm below Shaohai (anion).
  Interventions: Other: Shaohai session

INTERVENTIONS:
Other: sham electroacupuncture (EA) session — The stainless steels acupuncture needles inserted into the subcutaneous layer of Zusanli (cathode) and Shangjuxu acupints (anion) , and the needles connected to EA stimulator, but no electric discharge for 30 min.
  Arms: sham electroacupuncture (EA) session
Other: Zusanli session — The acupuncture needles inserted into Zusanli (cathode) and Shangjuxu acupoints (anion), and twisting obtain qi, and the needles then connected to EA stimulator, the frequency was 2 Hz, the duration was 30 min, and the intensity was visual slightly muscle contraction.
  Arms: Zusanli session
Other: Shaohai session — The methods were identical Zusanli group, but Shaohai acupoint (cathode), and 3 cm below Shaohai (anion).
  Arms: Shaohai session

SUMMARY:
The study on the relationship among meridian, acupoint and internal

DETAILED DESCRIPTION:
Meridian system is the pathway of transporting qi and blood, and that distributes all the body. Meridian system connects to internal visceral organs interior, and also connects to joints (or acupoint) exterior. The relationship among meridian, acupoints and internal visceral organs is still unclear. Therefore, the purpose of the present study was to investigate the relationship among meridian, acupoints and internal visceral organs. Total 33 subjects randomly finished three sessional studies as follows: 1) sham electroacupuncture (EA) session: the stainless steels acupuncture needles inserted into the subcutaneous layer of Zusanli (cathode) and Shangjuxu acupints (anion) , and the needles connected to EA stimulator, but no electric discharge for 30 min; 2) Zusanli session: the acupuncture needles inserted into Zusanli (cathode) and Shangjuxu acupoints (anion), and twisting obtain qi, and the needles then connected to EA stimulator, the frequency was 2 Hz, the duration was 30 min, and the intensity was visual slightly muscle contraction; 3) Shaohai session: the methods were identical Zusanli group, but Shaohai acupoint (cathode), and 3 cm below Shaohai (anion) . The major outcome measure was the changes of the percentage of gastric slow wave and dysrhythmia in 30 min electrogastrogram recordings, and the changes of cardiac output and stroke volume in 30 min recordings. Secondary outcome measure was the changes of saliva, blood and urine metabolites.

The investigators predict the results of the present study can test and verify meridian theory of traditional Chinese Medicine, meridian system connects internal visceral organ interior, and connects joint (or acupoint) exterior.

ELIGIBILITY:
Inclusion Criteria:

1. Gender：male or female.
2. Age：from 20 years old (inclusive) to 50 years old (inclusive).
3. After detailed description of the entire research purpose or process, voluntarily participate in the study and sign the consent form.

Exclusion Criteria:

1. Cancer, congestive hear failured NYHA class>II, COPD attack.
2. History of esophagus and gastroduodenal surgery、Barrett's esophagus.
3. Can not accept acupuncture points stimulators.
4. Allergic to acupuncture needles.
5. Has a mental illness or is unable to cooperate with the researcher.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
electrogastrogram recordings | 30 minutes in duration.
  the changes of the percentage of gastric slow wave .
cardiac output | 30 minutes in duration.
  the changes of cardiac output .
cardiac output | 30 minutes in duration.
  the changes of stroke volume .

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University Hospital, Taichung, North District, Taiwan